CLINICAL TRIAL: NCT07353424
Title: A Multicenter Randomized Clinical Trial Compared With Standard Clinical Practice to Evaluate the Efficacy of a Polyphenol-rich Salicornia Extract in the Progression of Cognitive Decline in a Cohort of Patients With Lacunar Infarcts
Brief Title: A Multicenter Randomized Clinical Trial Compared With Standard Clinical Practice to Evaluate the Efficacy of a Polyphenol-rich Salicornia Extract in the Progression of Cognitive Decline in a Cohort of Patients With Lacunar Infarcts (SALACUNAR)
Acronym: SALACUNAR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación Pública Andaluza para la gestión de la Investigación en Sevilla (Other)
Collaborators: Joan Montaner Villalonga (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SALACUNAR (LACI-2-polyphenols)
Record Dates: First submitted 2025-11-20; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Lacunar Stroke
Keywords: attack; food supplement; cognition
MeSH Terms: conditions — Stroke, Lacunar

STUDY DESIGN:
Intervention Model Description: Mulcenter, randomized, parallel-group, pilot trial aimed at evaluating the effect of the administration of a food supplement based on of a dietary supplement based on salicornia extracts in patients with cerebral small vessel disease patients with cerebral small vessel disease recruited in 15 SNS hospitals compared to the usual clinical clinical practice (PROBE).
Masking Description: Statistical analysis of data
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental): Food supplement to be taken once a day.
  Interventions: Dietary Supplement: B-salicornia
- Clinical practice (No Intervention): Without intervention

INTERVENTIONS:
Dietary Supplement: B-salicornia — Dietary supplement based on halophyte plant extracts (experimental) plus regular medical treatment. Dosage: once daily. Duration of study: 6 months.
  Arms: Treatment

SUMMARY:
SALACUNAR (LACI-2-polyphenols) is a multi-center randomized controlled trial (RCT) to evaluate the effect of a polyphenol-rich supplement on small vessel neurovascular disease. Specifically, the compound to be tested is a dietary supplement based on Salicornia extract and B vitamins (B-salicornia), which in previous studies has demonstrated a good safety profile and consistent effects in reducing homocysteine levels and improving cognitive outcomes (MOCA) in patients with lacunar infarcts. This has been used to calculate the sample size based on these endpoints. Considering an intragroup variability of the treatment groups (sigma) of 6.07, and accepting an alpha risk of 0.05, a sample of 150 patients per group would achieve a 1-beta statistical power greater than 0.8 in a two-tailed test for differences between means of at least two points on the MOCA scale.

Three hundred patients with lacunar infarcts diagnosed within the last year and confirmed by MRI performed as part of routine clinical practice will be included.

We will administer 500 mg/24 h of the dietary supplement B-Salicornia for six months (or the control group will be managed according to routine clinical practice) following a PROBE design.

Routine blood tests will be performed pre- and post-treatment, with routine vascular parameters such as lipids and homocysteine, as well as baseline and six-month assessments of neuropsychological and gait scales.

ELIGIBILITY:
Inclusion Criteria:

- Patients with lacunar ischemic stroke, confirmed by cranial magnetic resonance imaging performed within the year prior to inclusion, who have an mRS of 3 or less at the time of inclusion will be included (independent patients or those who require assistance with walking). The inclusion age will be between 40 and 90 years.

Exclusion Criteria:

* Consumption of vitamin supplements or polyphenol supplements within 30 days prior to inclusion
* Hyperthyroidism
* mRS >3, serious illness, or expected life expectancy <12 months
* Dysphagia preventing intake of the study capsules
* Allergies or intolerance to halophytes
* Pregnant or breastfeeding
* Active neoplasia
* Participation in another study

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Six-minute walk test (6MWT) | 6 months
  To evaluate changes in walking performance in patients who took the supplement compared to patients who followed standard clinical practice.
Neuropsychological questionnaires: Montreal Cognitive Assessment (MOCA) | 6 months
  Assess possible improvements in cognitive function in patients taking the supplement versus patients following standard clinical practice.
Blood laboratory parameters (homocysteine µmol/L). | 6 months
  Measurement of changes in blood tests in patients taking the dietary supplement compared to patients following standard clinical practice.
Morisky-Green test count of returned treatment capsules. | 6 months
  Confirm adequate adherence to dietary supplementation.
Severity of the adverse event. | 6 months
  - Mild: No antidote or treatment required; brief hospitalisation. - MODERATE: Treatment modification required (e.g., dose change, addition of another drug), but discontinuation of the drug is not essential; prolonged administration of the drug is not essential; prolonged hospitalisation or treatment may be necessary, or specific hospitalisation or treatment may be necessary. - SEVERE: The adverse drug reaction is life-threatening and requires discontinuation of the drug. Drug administration should be discontinued and specific treatment instituted. - FATAL: An adverse drug reaction may directly or indirectly contribute to the death of the patient.

SECONDARY OUTCOMES:
Blood laboratory parameters (total cholesterol mg/dl). | 6 months
  Measurement of changes in blood tests in patients taking the dietary supplement compared to patients following standard clinical practice.
Blood laboratory parameters (Low density lipoprotein cholesterol mg/dl). | 6 months
  Measurement of changes in blood tests in patients taking the dietary supplement compared to patients following standard clinical practice.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario Virgen Macarena, Seville, Spain